CLINICAL TRIAL: NCT00224458
Title: Combination of Efavirenz & Truvada (COMET Study): Phase 4 Evaluation of Switching Twice Daily Combivir to Once-Daily Regimen Co-Formulated Truvada in Virologically Suppressed HIV Infected Patients Taking Efavirenz.
Brief Title: Combination of Efavirenz and Truvada - COMET Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: John Flaherty, Director, Medical Affairs, Gilead Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-164-0107
Record Dates: First submitted 2005-09-19; First posted 2005-09-23 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-02

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz

INTERVENTIONS:
Drug: Truvada
Drug: efavirenz

SUMMARY:
To characterize the risks (safety and tolerability), effectiveness (continued viral load suppression and CD4 changes), and benefits (safety, tolerability, adherence, general satisfaction with the treatment regimen and QoL), of switching from a Combivir (BID) / efavirenz (QD) regimen to an all QD regimen of Truvada/efavirenz.

DETAILED DESCRIPTION:
The objectives of this study are to characterize the risks (safety and tolerability), effectiveness (continued viral load suppression and CD4 changes), and benefits (safety, tolerability, adherence, general satisfaction with the treatment regimen and QoL), of switching from a Combivir (BID) / efavirenz (QD) regimen to an all QD regimen of Truvada/efavirenz.

ELIGIBILITY:
Inclusion Criteria:

* Adult (greater than 18 years) male or non-pregnant female HIV-1 infected patients regardless of race or ethnicity.
* On a stable antiretroviral regimen consisting of efavirenz QD and Combivir BID for greater than 8 weeks.
* Plasma HIV 1 RNA less than 400 copies/mL (Roche Amplicor HIV 1 Monitor Test Version 1.5 Ultrasensitive method).
* Currently experiencing adverse clinical or laboratory effects associated with Combivir and/or who might benefit from a simplified, once-daily antiretroviral treatment regimen regardless of Combivir tolerability status.
* Adequate renal function defined as a calculated creatinine clearance (CLCr) greater than or equal to 50 mL/min according to the Cockcroft-Gault formula:

Male: (140 - age in years) x (wt in kg) divided by 72 x (serum creatinine in mg/dL) = CLCr (mL/min.

Female: (140 - age in years) x(wt in kg) divided by 72 x (serum creatinine in mg/dL) x 0.85 = CLCr (mL/min).

* Negative serum pregnancy test (females of childbearing potential only).
* Willingness to use effective contraception (such as barrier or coil methods) by both males and females while on study drug and for 30 days following study drug completion.
* Life expectancy less than 1 year.
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Exclusion Criteria:

* A new AIDS defining condition diagnosed (with the exception of CD4 criteria) within 30 days of baseline.
* Clinically significant laboratory values that would preclude prescribing antiretroviral therapy, in the opinion of the investigator.
* Receiving on-going therapy with any of the following (administration of any of the following medications must be discontinued at least 30 days prior to the Baseline visit and for the duration of the study period):
* Nephrotoxic agents (aminoglycoside antibiotics, IV amphotericin B, cidofovir, cisplatin, foscarnet, IV pentamidine, other agents with significant nephrotoxic potential):

  * Adefovir dipivoxil
  * Probenecid
  * Systemic chemotherapeutic agents (i.e., cancer treatment medications)
  * Systemic corticosteroids
  * Interleukin 2 (IL 2)
  * Investigational agents (except upon approval by Gilead).
* Drugs that interact with efavirenz:

  * dihydroergotamine
  * ergotamine
  * ergonovine
  * methylergonovine
  * midazolam
  * triazolam
  * cisapride
  * rifampin
* Pregnant or lactating patients.
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with patient adherence.
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Patients with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and are not anticipated to require systemic therapy during the study.
* Active, serious infections (other than HIV 1 infection) requiring parenteral antibiotic therapy within 15 days prior to screening.
* Prior history of significant renal or bone disease.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-09; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To characterize the risks (safety and tolerability), effectiveness (continued viral load suppression and CD4 changes), and benefits (safety, tolerability, adherence, general satisfaction with the treatment regimen and QoL)

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences

REFERENCES:
- [Derived] DeJesus E, Ruane P, McDonald C, Garcia F, Sharma S, Corales R, Ravishankar J, Khanlou H, Shamblaw D, Ecker J, Ebrahimi R, Flaherty J; COMET Study Team. Impact of switching virologically suppressed, HIV-1-infected patients from twice-daily fixed-dose zidovudine/lamivudine to once-daily fixed-dose tenofovir disoproxil fumarate/emtricitabine. HIV Clin Trials. 2008 Mar-Apr;9(2):103-14. doi: 10.1310/hct0902-103. PMID 18474495
- See also: Gilead Website — http://www.gilead.com
- See also: Truvada Website — http://www.truvada.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-US-164-0107_synopsis.pdf